CLINICAL TRIAL: NCT07085897
Title: Efficacy of an Integrated Growth Mindset Intervention on Reducing Anxiety for Practicum Training Among Students in the Allied Health Professions: Study Protocol for a Two-Arm Randomised Controlled Trial
Brief Title: Web-based Single-session Growth Mindset Intervention for Allied Health Practicum Trainees to Reduce Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSEARS20250608002
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) (Experimental): The intervention is structured into three video-and-exercise sessions. Part one focuses on students' mindsets in coping with practicum-related challenges and their attitudes towards setbacks, encouraging them to shift from a 'fear-of-failure' mindset to a 'failure-is-enhancing' mindset. Part two introduces the nature and concept of neuroplasticity to promote students' understanding of effective learning. Part three centers on providing guidance for students on strategies to cope with stress and emotional turbulence with growth mindset regarding emotion.
  Interventions: Behavioral: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) for allied health practicum trainees
- Training-as-usual group (No Intervention): The training-as-usual group will continue the regular practicum training.

INTERVENTIONS:
Behavioral: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE) for allied health practicum trainees — The intervention is structured into three video-and-exercise sessions. Part one focuses on students' mindsets in coping with practicum-related challenges and their attitudes towards setbacks, encouraging them to shift from a 'fear-of-failure' mindset to a 'failure-is-enhancing' mindset. Part two introduces the nature and concept of neuroplasticity to promote students' understanding of effective learning. Part three centers on providing guidance for students on strategies to cope with stress and emotional turbulence with growth mindset regarding emotion.
  Arms: Web-based Single-session Intervention of Mindset on Intelligence, Failure, and Emotion (We-SMILE)

SUMMARY:
Practicum is a critical component of professional training, offering essential experiential learning opportunities that support the development of future practitioners. However, existing research indicates that practicum can be particularly challenging for allied health students, who must navigate both academic learning adjustments and complex healthcare environments. Emerging evidence also highlights the potential value of low-intensity, self-guided interventions in enhancing practicum trainees' psychological preparedness. Based on the findings, this present project adapts an integrated intervention-the Web-based Single-Session Intervention on Mindset regarding Intelligence, Failure, and Emotion (We-SMILE)-specifically for practicum students in allied health professions and examines its efficacy to adjust their mindsets and manage practicum-related challenges more effectively.

Using a two-arm randomised controlled trial, the proposed study will examine the efficacy of We-SMILE for allied health practicum trainees in reducing anxiety, as well as improving perceived stress, performance anxiety, practicum-related concerns, psychological status, learning orientation, confidence, resilient coping, and time management.

Students commencing their practicums will be recruited from allied health programmes and randomly assigned to either existing pre-practicum training plus intervention or the training-as-usual control group. Participants will be assessed at three time-points: baseline before intervention (T1), two weeks post-intervention (T2) and two months post-intervention (T3). The intention-to-treat principle and linear-regression-based maximum likelihood multi-level models will be used for data analysis.

Feasibility and Potential: This project brings together experts in mindset research, fieldwork coordinators, and programme leaders, ensuring the feasibility of the study. It will not only generate evidence on the adapted We-SMILE intervention for allied health practicum trainees but also offer a scalable and accessible model for enhancing the well-being of trainees in other healthcare and helping professions.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in allied health programmes who are about to commence their practicums or have recently entered practicum.

Exclusion Criteria:

* (1) do not consent to participate, (2) cannot concentrate for at least 45 minutes to complete the intervention and questionnaires, (3) have a disability or serious physical or mental illness resulting in poor condition, and (4) do not participate in the practicum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety related to practicum | Baseline, 2-week and 8-week follow-ups
  Anxiety related to practicum will be measured by four items, including "level of anxiety about starting the practicum", "how much your anxiety will interfere with their learning", "how prepared you are for the practicum" and "how excited you are to participate in the practicum". Each statement will be rated on a 10-point Likert scale, ranging from 1=completely not anxious, very small, completely unprepared, and completely unexcited to 10=extremely anxious, very great, perfectly prepared, and extremely excited.

SECONDARY OUTCOMES:
Psychological states | Baseline, 2-week and 8-week follow-ups
  Psychological states will be assessed by the Depression, Anxiety and Stress Scale-8 Items (DASS-8) is a set of three self-report scales designed to measure the psychological states of depression, anxiety and stress. Each of the depression and anxiety sub-scales of the DASS-8 contain 3 items while the stress sub-scale contains 2 items. Each item can be scored from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time).
Performance anxiety | Baseline, 2-week and 8-week follow-ups
  Performance anxiety will be examined by the sub-scale of cognitive anxiety from the Performance Test Anxiety questionnaire (PTA). Respondents indicated how they were thinking and feeling about their practicum (using a 5-point scale on which 1=totally disagree and 5=totally agree) in response to the items.
Learning orientation | Baseline, 2-week and 8-week follow-ups
  Learning orientation will be assessed by five items (e.g., "I like to learn new knowledge in practicums."). Each item will be rated by a five-point Likert scale from 1=strongly disagree to 5=strongly agree.
Confidence | Baseline, 2-week and 8-week follow-ups
  Confidence will be assessed by a six-item self-developed scale. Items generated from interviews with practicum students, such as "I am confident that I can listen to comments from supervisors/colleagues/service users with an open mind." and "I am confident that I can manage my time well and cope with my practicum work and schoolwork at the same time.". Each item needs to be rated from 1=strongly disagree to 5=strongly agree.
Resilient Coping | Baseline, 2-week and 8-week follow-ups
  Resilient Coping will be measured by a self-report four-item Brief Resilient Coping Scale (BRCS). Items will be scored from 1 (Does not describe me at all) to 5 (Describe me very well). A sample item is "I look for creative ways to alter difficult situations".
Perceived stress | Baseline, 2-week and 8-week follow-ups
  Stress will be examined by the Perceived Stress Scale-4 items (PSS-4). It measures the degree to which situations in one's life over the past month are appraised as stressful. Each item will be scored from 0 (Never) to 4 (Very often). Total score is determined by adding together the scores of each of the four items. Questions 2 and 3 are reverse coded.
Practicum-related concerns | Baseline, 2-week and 8-week follow-ups
  Practicum-related concerns will be assessed using a self-developed six-item scale designed to reflect the concerns of allied health students.
Time management | Baseline, 2-week and 8-week follow-ups
  Time management will be assessed using the 'Setting Goals and Priorities' sub scale of the Time Management Behavior (TMB) Scale, which includes ten items. Each item is rated on a 5-point Likert scale ranging from 1 (seldom true) to 5 (very often true).

IPD SHARING:
Plan to Share IPD: Undecided